CLINICAL TRIAL: NCT02422030
Title: A Randomized, Open-label, Multiple Dosing, 3-way Crossover Study to Evaluate the Drug-drug Interaction Between Atorvastatin and Fenofibric Acid in Healthy Male Volunteers
Brief Title: CKD-337(2) Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146DDI14030
Record Dates: First submitted 2015-03-25; First posted 2015-04-21 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Male Volunteers
MeSH Terms: interventions — Atorvastatin; Fenofibrate; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group1: TreatmentA+TreatmentB+TreatmentC (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg
- Group2: TreatmentC+TreatmentA+TreatmentB (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg
- Group3: TreatmentB+TreatmentC+TreatmentA (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg
- Group4: TreatmentC+TreatmentB+TreatmentA (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg
- Group5: TreatmentB+TreatmentA+TreatmentC (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg
- Group6: TreatmentA+TreatmentC+TreatmentB (Experimental): TreatmentA: Atorvastatin 40m*1T/day, TreatmentB: Fenofibric acid 135mg*1Cap/day, TreatmentC: Atorvastatin 40m*1T/day and Fenofibric acid 135mg*1Cap/day. Each treatment period was separated by a washout period of at least 8days.
  Interventions: Drug: Lipitor Tab. 40mg; Drug: Trilipix 135mg

INTERVENTIONS:
Drug: Lipitor Tab. 40mg
  Other Names: Atorvastatin 40mg
Drug: Trilipix 135mg
  Other Names: Fenofibric acid 135mg

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic interaction between Atorvastatin and Fenofibric acid.

DETAILED DESCRIPTION:
This study is a randomized, open-label, multiple dosing, 3-way crossover design to evaluate the drug-drug interaction between Atorvastatin (Lipitor) and Fenofibric (Trilipix) acid in healthy male subjects. Subjects will receive repeated dose of Atorvastatin (40mg*1Tab/day) or Fenofibric acid (135mg*1Cap/day) or Atorvastatin (40mg*1Tab/day)/Fenofibric acid (135mg*1Cap/day). Each treatment period was separated by a washout period of at least 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man older than 19 years at the time of screening.
* BMI more than 17.5kg / m2 and less than 30.5kg / m2 and weight more than 55kg
* Subject without congenital or chronic diseases and no psychotic symptoms or findings from the medical examination.
* Suitable subject who is determined by laboratory tests such as hematology tests, blood chemistry, urinalysis test according to the characteristics of the drug and screening tests such as ECG test.
* Subject who fully understand the clinical trials after in-depth explanation given prior to the clinical study, decided to join the clinical trials by their will and signed consent form which approved by Chonbuk National University Hospital IRB.
* Subjects who are able to comply with all scheduled visits, laboratory tests and other procedures.

Exclusion Criteria:

1. Subject who has a history of blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic diseases that is clinically significant (Except untreated asymptomatic seasonal allergies at the time of administration)
2. Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption.
3. Showing the value that corresponds to following laboratory parameters: AST or AST or CK > 2* upper limit of normal range.
4. Alcohol > 210g/week, within 6 months prior to the screening.
5. Taking the medication involved in other clinical trials within two months before the first dose medication characters.
6. Sitting Systolic Blood Pressure ≥ 140 mmHg, Diastolic Blood Pressure ≥ 90 mmHg at the time of screening.
7. History of alcohol or drug abuse, within 1 year
8. Subjects who treated with metabolizing enzyme inducers or inhibitors such as barbitals within 30days prior to the first dosing.
9. Smoker (> 20cigarettes/day)
10. Subjects who takes ETC or OTC medicine within 10days before the first IP administration.
11. Subject who done the whole blood donation within two months or component blood donation within 1 month within 1 month prior to the first dosing.
12. Subject who can increase risk due to clinical test and administration of drugs or has Severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
13. Subject with serious history of hypersensitivity or allergy to investigational product.
14. Active liver disease.
15. Muscle disease.
16. Subject with genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption.
17. Patients with severe hepatic impairment or Gallbladder Disease.
18. Patients with moderate to severe renal impairment.
19. Patients experienced allergy or phototoxicity during treatment with fibrate or ketoprofen.
20. Subjects who is not able to comply with guidelines described in the protocol.
21. Subjects who is determined by investigator's decision as unsuitable for clinical trial participation.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2015-03-22 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Atorvastatin and Fenofibric acid AUCτ | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points
Atorvastatin and Fenofibric acid Css,max | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points

SECONDARY OUTCOMES:
Atorvastatin and Fenofibric acid Css,min | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points
Atorvastatin and Fenofibric acid Css,av | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points
2-hydroxyatorvastatin AUCτ | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points
2-hydroxyatorvastatin Css,max | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours post-dose, an expected average of 6weeks
  1D~7D 19points, 1D~7D 18points, 1D~7D 20points

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Deokjin-gu, Jeonju-si, Jeollabuk-do, South Korea